CLINICAL TRIAL: NCT02334761
Title: Biopsies in Oncology - Prospective Study of Impact on Patient's Quality of Life.
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: BIOPSy
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Pathology
Keywords: Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Over the past decade the paradigm of care in oncology has evolved with the advent of personalized medicine. Yet, despite this exciting prospect, there are currently only a few disease subtypes where therapeutic approaches with proven benefit exist such as EGFR (Epidermal Growth Factor Receptor) targeted therapies in EGFR-mutant lung tumours. With the increasing number of novel molecularly targeted agents available, the importance of building our understanding of cancer biology is critical.

Challenges to implement personalized medicine include the limitations of molecular testing, tumour heterogeneity and molecular evolution, costs, and the quality and morbidity associated with tumour biopsies. Sequential biopsies are essential to better understand biological markers of response and resistance, and identify predictive or prognostic markers. Despite the scientific rationale for biopsies, incorporating them into practice can be challenging, as in many cases there is no direct advantage to the patient. This project aims to understand the effect of research biopsies on the patient. The Investigator hypothesize by learning more and gaining a better appreciation of the impact on the patient, Investigators will increase the likelihood of achieving serial biopsies.

The ability to obtain serial biopsies is dependent on the patient's experience. To understand the clonal progression of cancer and validate predictive and prognostic markers of response, studies now target biopsies both at enrollment and at progression. As Investigators strive to achieve this, improving our understanding of the patient's experience will help us identify factors that positively and negatively impact on patient participation and influence the probability of successfully obtaining sequential samples.

DETAILED DESCRIPTION:
Both primary and secondary objectives will be assessed in a questionnaire. Primary Objectives To assess the impact of research biopsies on patients quality of life.

Secondary Objectives To assess the impact of diagnostic biopsies on quality of life in comparison to research biopsies.

To assess the true complication rates associated with biopsies. To compare types of biopsies - surgical versus radiological with respect to implications on quality of life.

To assess the individual potentially modifiable factors of reason for biopsy; perceived risk; perceived benefit; wait time for biopsy; wait time for results; complications; and altruism and association with anxiety.

To determine which factors are associated with a higher and lower likelihood of achieving serial biopsies.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

Patient must be ≥18 years old. ECOG (Eastern Cooperative Oncology Group) performance status ≤2 (Karnofsky ≥60%).

Life expectancy of greater than 3 months Must be undergoing a biopsy for research or diagnostic purposes. Have a diagnosis of malignancy or an assumed diagnosis of malignancy in patients where the biopsy is being performed for diagnostic purposes.

Able to complete questionnaires independently. Ability to understand and the willingness to sign a written informed consent document.

Both men and women of all races and ethnic groups are eligible for this trial. Verbal translation will be available for the consent and assistance with the questionnaires. If language is a second language or the patient is unable to read the questionnaire for any reason a family member may assist with the questionnaires.

Exclusion Criteria:

Patients who do not have a biopsy scheduled and performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient must be 18 years or older with a life expectancy of greater than 3 months. The patient must be undergoing a biopsy for research or diagnostic purposes with a diagnosis of malignancy or an assumed diagnosis of malignancy. The patient must be able to complete the questionnaires independently.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the impact of research biopsies on patients quality of life. | 6-8 months

SECONDARY OUTCOMES:
To assess the impact of diagnostic biopsies on quality of life in comparison to research biopsies | at minimum: 6 months
To assess the true complication rates associated with biopsies | at minimum: 6 months
To compare types of biopsies - surgical versus radiological with respect to implications on quality of life | at minimum: 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Madariaga A, Bhat G, Wilson MK, Li X, Cyriac S, Bowering V, Hunt W, Gutierrez D, Bonilla L, Kasherman L, McMullen M, Wang L, Ghai S, Dhani NC, Oza AM, Lheureux S. Research biopsies in patients with gynecologic cancers: patient-reported outcomes, perceptions, and preferences. Am J Obstet Gynecol. 2021 Dec;225(6):658.e1-658.e9. doi: 10.1016/j.ajog.2021.06.071. Epub 2021 Jun 23. PMID 34174204